CLINICAL TRIAL: NCT04080180
Title: Testing the Effects of Contingency Management and Behavioral Economics on Buprenorphine-Naloxone Treatment Adherence Using a Sequential Multiple Assignment Randomized Trial (SMART) Design
Brief Title: SMART Trial for Buprenorphine-Naloxone Medication Assisted Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Derefinko, PhD (Other)
Collaborators: University of Memphis (Other); University of New Mexico (Other); University of Tennessee (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Karen Derefinko, PhD, Assistant Professor, University of Tennessee
Organization: University of Tennessee (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 19-06690-FB; 1R61AT010604-01 (NIH)
Record Dates: First submitted 2019-08-16; First posted 2019-09-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Opioid-use Disorder
Keywords: opioid use disorder; buprenorphine; treatment adherence
MeSH Terms: conditions — Opioid-Related Disorders; Treatment Adherence and Compliance | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: In stage 1, participants are individually randomized (1:1) to BSM or CM. At the end of stage 1, adherent buprenorphine-naloxone participants remain in their respective intervention group during phase 2 (maintenance phase of same approach), whereas non-adherent participants are randomized (individually and 1:1) to either switch or add the respective other intervention in this part-factorial SMART. Our primary outcome is buprenorphine-naloxone adherence by the end of stage 2. This sequential randomization based on past treatment success assures that the assigned treatment option at any point in time is independent of future potential outcomes and only conditional on the subject's history, i.e., the sequential ignorable treatment assumption is satisfied by design,108 in sharp distinction to observational data where patients chose to switch/add or not to switch/add and where this assumption remains untestable.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Contingency Management (CM) (Active Comparator): CM is a behavioral method that employs external rewards for target behavior. Participants will receive gift cards for adhering to treatment (attending physician visits and being adherent to buprenorphine-naloxone) for their first 4 clinic visits.
  Interventions: Behavioral: Contingency Management
- Brief Motivational Interviewing + Substance Free Activities + Mindfulness (BSM) (Active Comparator): Participants will receive the BSM intervention at 4 timepoints.
  Interventions: Behavioral: Brief Motivational Interviewing + Substance Free Activities + Mindfulness
- BSM+CM (Active Comparator): BSM+CM is a combination of the two other arms. Participants may be randomized to this arm only in stage 2 of the SMART design.
  Interventions: Behavioral: Contingency Management; Behavioral: Brief Motivational Interviewing + Substance Free Activities + Mindfulness

INTERVENTIONS:
Behavioral: Contingency Management — Contingency management (CM) is a behavioral method that employs external rewards for target behavior. For this study, participants will receive gift cards for adhering to Medication-Assisted Treatment (attending physician visits and adhering to buprenorphine-naloxone as determined by urine toxicology panel) during their first four visits while randomized to this condition. Participants will draw a gift card from a fishbowl each visit they are adherent. Gift cards range from $25-$100.
  Other Names: CM
  Arms: BSM+CM; Contingency Management (CM)
Behavioral: Brief Motivational Interviewing + Substance Free Activities + Mindfulness — Brief Motivational Interviewing + Substance Free Activities + Mindfulness (BSM) is an intervention that uses Motivational Interviewing and Behavioral Economics strategies to increase the salience of delayed rewards by eliciting personal goals, developing opioid-free activities, and engaging in reward bundling and episodic future thinking. Participants will be offered a menu of substance free activities that has been developed in pilot work. Activities will be discussed, and participants will be asked to engage in selected activities as homework. Engagement in substance free activities will be assessed at each subsequent visit. Mindfulness components will also be included in the intervention.
  Other Names: BSM
  Arms: BSM+CM; Brief Motivational Interviewing + Substance Free Activities + Mindfulness (BSM)

SUMMARY:
The purpose of this study is to compare the effectiveness of two different interventions for medication-assisted treatment (MAT) adherence: Contingency Management (CM) and Brief Motivational Interviewing + Substance Free Activities + Mindfulness (BSM).

DETAILED DESCRIPTION:
The investigators seek to compare the effectiveness of these two different interventions for MAT adherence by first refining and piloting CM and BSM adherence approaches, then conducting a Sequential Multiple Assignment Randomized Trial (SMART) to assess sequential, individual, and combined effects across MAT initiation and maintenance.

In order to tailor treatment to individual's needs, the study will follow a sequential multiple assignment randomized trial (SMART) design: In stage 1, participants are individually randomized (1:1) to BSM or CM. Adherent buprenorphine-naloxone participants complete treatment in the arm they were originally assigned to, but non-adherent participants are re-randomized (1:1) to either switch to the other intervention or add the other intervention in this part-factorial SMART.

ELIGIBILITY:
Inclusion Criteria:

* Present with symptoms of Opioid Use Disorder
* Eligible of receipt of buprenorphine-naloxone medication as determined by Study Doctor
* Access to a telephone

Exclusion Criteria:

* Under 18 years old
* Unable to understand spoken English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Medication-Assisted Treatment (MAT) Adherence | through study completion, an average of 8 months
  Number of visits where participant attends physician appointment and drug screen results are buprenorphine-positive.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that a cleaned data set of study-specific data will be provided within two years following the completion of the study for the data archive and this data set would be made public. Confidentiality of individual participants would be maintained with all releases of data. The final study analytical database would be processed according to HIPAA definitions for public data sharing. Documentation would be provided along with the data sharing file that includes but is not limited to: data dictionary, data codebook, valid variable ranges (where provided), the protocol, procedure and operational manuals, intervention manual or programs and any electronic versions of any paper forms that were used in data collection.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within two years of study completion.

REFERENCES:
- [Derived] Peter SC, Murphy JG, Witkiewitz K, Hand SB, Thomas F, Johnson KC, Cowan R, Harris M, Derefinko KJ. Use of a sequential multiple assignment randomized trial to test contingency management and an integrated behavioral economic and mindfulness intervention for buprenorphine-naloxone medication adherence for opioid use disorder. Trials. 2023 Mar 29;24(1):237. doi: 10.1186/s13063-023-07102-9. PMID 36991453

DOCUMENTS (1):
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04080180/ICF_000.pdf